CLINICAL TRIAL: NCT00173238
Title: The Study of Human Atherosclerosis by Polarization-Sensitive Optical Coherence Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700533
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-06

CONDITIONS: Pathological Conditions, Anatomical
Keywords: atherosclerosis; optical coherence tomography; polarization; phase retardation; birefringence
MeSH Terms: conditions — Pathological Conditions, Anatomical; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Atherosclerosis is unquestionably the leading cause of morbidity and mortality in developed countries, and the world-wide importance of acute vascular syndromes is increasing. Rupture of atherosclerotic plaque has been identified as the proximate event in the majority of cases of acute ischemic syndromes. Therefore, modalities capable of characterizing the atherosclerotic lesion may be helpful in understanding its natural history and detecting lesions with high risk for acute events.

Optical coherence tomography (OCT) is a powerful tool capable of tomographic imaging based on low coherence interferometry. It is analogous to ultrasound imaging except that it uses infrared light instead of sound. Polarization-sensitive optical coherence tomography (PS-OCT) combines the advantages of OCT with additional image contrast of the sample. The added contrast is based on the ability of PS-OCT to detect the birefringent properties of a sample (phase retardation and fast-axis orientation) simultaneously.

The goals of this project are: 1) to examine whether PS-OCT is an acceptable tool for the characterization of typical plaque constituents; and 2) to explain the correlation between birefringence and forming or rupture of a plaque; and 3) to establish a quantitative PS-OCT image criteria for atherosclerotic plaque characterization in vitro.

DETAILED DESCRIPTION:
Optical Coherence Tomography (OCT) is a promising new class of diagnostic medical imaging technology that utilizes advanced photonics and fiber optics to obtain images and tissue characterization on a scale never before possible within the human body. OCT combines the principles of ultrasound with the imaging performance of a microscope and a form factor that is familiar to clinicians. Whereas ultrasound produces images from backscattered sound "echoes," OCT uses infrared light waves that reflect off the internal microstructure within the biological tissues.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplantation, atherosclerosis

Exclusion Criteria:

* Infection

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5
Dates: Start 2005-06; Study Completion 2008-06

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Kuan Chou, MD.,PhD, Principal Investigator — National Taiwan University Hospital,Taipei.Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan